CLINICAL TRIAL: NCT06818435
Title: Portuguese Registry With Meril Myval THV Series - MyPORTuVal Registry
Acronym: MyPORTuVal
Status: Recruiting | Type: Observational
Sponsor: Portuguese Association of Interventional Cardiology (Other)
Collaborators: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MyPTVal-1
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Stenosis; TAVI(Transcatheter Aortic Valve Implantation)
Keywords: MyPORTuVal; TAVI; Portuguese TAVI Registry
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Myval THV series — Transcatheter Aortic Valve Implantation

SUMMARY:
A prospective, single-arm, multi-centre registry to evaluate the safety and performance of Myval THV series using Transcatheter Aortic Valve Implantation (TAVI) procedure in patients with symptomatic severe native aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over the age of 18 years with symptomatic aortic stenosis (severe AS), intended to perform TAVI procedure using Myval THV series as assessed by Heart Team.
2. Patient has provided written informed consent as approved by the Ethics Committee (EC)
3. Patient is willing to undergo all registry procedures and follow-up requirements

Exclusion Criteria:

1. Patients with hyper sensitivity or allergy to aspirin, heparin, clopidogrel, ticlopidine, cobalt, nickel, chromium, molybdenum or any contrast media.
2. Ongoing infective endocarditis or any similar infection.
3. Pregnant or lactating females.
4. Liver failure (Child-Pugh Class B or C)
5. Patient is currently participating in another clinical investigation where the primary endpoint has not been achieved.
6. Any condition, which in the investigator opinion, would preclude safe participation of the patient in the Registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic severe native aortic valve stenosis who underwent TAVI using Myval THV series as assessed by Heart Team and Investigator.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Safety of Myval valve and TAVI procedure | 30 days
  Composite of:
  * All-cause mortality
  * All stroke
  * Acute kidney injury (stage 2, 3 and 4)
  * Bleeding (Type 3 and 4)
  * Moderate or severe paravalvular leak
  * Major vascular complications
  * Conduction disturbances resulting in new permanent pacemaker implantation

SECONDARY OUTCOMES:
Safety and Performance of Myval valve and TAVI procedure | 30 days and 12 Months
  1. All-cause mortality (cardiac and non-cardiac)
  2. All stroke
  3. Acute Kidney Injury (AKI) System-Stage 2, 3 and 4
  4. Moderate or severe paravalvular leak
  5. Conduction disturbances and Arrythmias
  6. New permanent pacemaker implantation
  7. Major vascular complications
  8. Vascular and access related complications
  9. Echocardiography measurements
  10. Procedure-related assessments
  11. New York Heart Association (NYHA) Functional Classification
  12. Re-Hospitalization
  13. Bleeding (Type 3 and 4)
  14. Myocardial Infarction
  15. Length of index hospital stay
  16. Cardiac structural complications
  17. Aortic bioprosthetic valve dysfunction
  18. Bioprosthetic valve deterioration
  19. Conversion to open surgery
  20. Unplanned use of mechanical circulatory support
  21. Implantation of multiple (>1) transcatheter valves during the index hospitalization
  22. Valve malposition
  23. Technical success
  24. Device success
  25. Early safety

CONTACTS AND LOCATIONS:
Overall Officials: Rui Campante Teles, Prof. Dr., Study Chair — Unidade Local de Saúde de Lisboa Ocidental, E.P.E. - Hospital de Santa Cruz
Locations (6):
- Portugal (6):
  - Unidade Local de Saúde do Lisboa Ocidental E.P.E. - Hospital Santa Cruz, Carnaxide
  - Unidade Local de Saúde de Coimbra, Coimbra
  - Unidade Local de Saúde Alentejo Central E.P.E. - Hospital Espírito Santo, Evora
  - Unidade Local de Saúde de São José E.P.E. - Hospital Santa Marta, Lisbon
  - Unidade Local de Saúde de Santa Maria, E.P.E. - Hospital de Santa Maria, Lisbon
  - Unidade Local de São João E.P.E., Porto

IPD SHARING:
Plan to Share IPD: No